CLINICAL TRIAL: NCT07271875
Title: Effect of Neuromuscular Reversal With Neostigmine/Atropine Versus Sugammadex on Postoperative Gastrointestinal Function Recovery Following Colorectal Surgery
Brief Title: Neuromuscular Blocking Agents on Gastrointestinal Function Following Colorectal Surgery
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Chong Lei, MD & phD, Professor. MD &phD, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KY20252236
Record Dates: First submitted 2025-09-22; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Gastrointestinal Dysfunction (POGD); Postoperative Ileus; Colorectal Surgery
MeSH Terms: interventions — Neostigmine; Atropine; Sugammadex

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Statisticians are also masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sugammadex group (Experimental): Sugammadex 2 mg/kg administered after surgery
  Interventions: Drug: Sugammadex
- Neostigmine group (Active Comparator): Neostigmine 30 μg/kg + Atropine 15 μg/kg administered after surgery
  Interventions: Drug: Neostigmine + Atropine

INTERVENTIONS:
Drug: Neostigmine + Atropine — Participants received Neostigmine 30 μg/kg + Atropine 15 μg/kg after surgery once a train-of-four ratio of 0.9 and sufficient spontaneous breathing were confirmed.
  Arms: Neostigmine group
Drug: Sugammadex — Participants received sugammadex 2 mg/kg after surgery once a train-of-four ratio of 0.9 and sufficient spontaneous breathing were confirmed.
  Arms: Sugammadex group

SUMMARY:
This study is a clinical research project conducted at Xijing Hospital to compare the effects of two different neuromuscular blockade reversal strategies on the recovery of gastrointestinal (GI) function after colorectal surgery.

Many patients experience slow recovery of bowel function after colorectal surgery, which can lead to discomfort, nausea, vomiting, and a longer hospital stay. This study investigates whether using one medication (sugammadex) to reverse muscle relaxants used during anesthesia leads to better and faster recovery of gastrointestinal function compared to a traditional combination of medications (neostigmine with atropine).

The study will include 560 adults scheduled for elective colorectal surgery. Participants will be randomly assigned to one of two groups to receive either:

Sugammadex (2 mg/kg), OR Neostigmine (30 μg/kg) + Atropine (15 μg/kg) The assigned study drug will be given by intravenous injection at the end of surgery, once measurements show the muscle relaxant is starting to wear off. The patients, surgeons, outcome assessors, and statisticians will be blinded.

The main goal is to see if more patients in one group recover their gastrointestinal function within 72 hours after surgery. Gastrointestinal recovery is strictly defined as both being able to tolerate food/drinks without significant nausea/vomiting AND having passed gas or had a bowel movement.

The study will also compare many other important outcomes between the groups, including:

1. Time to first passage of gas, first bowel movement, and first toleration of food.
2. Pain scores and opioid pain medication use.
3. Rates of nausea and vomiting.
4. Overall quality of recovery and patient satisfaction.
5. Length of hospital stay and total hospitalization costs.
6. Occurrence of complications within 30 days after surgery.
7. The safety of both reversal strategies will be closely monitored throughout the study by recording any adverse events.

This research aims to provide high-quality evidence to help anesthesiologists and surgeons choose the best method to reverse muscle relaxation, potentially leading to faster recovery, fewer complications, and a better overall experience for patients undergoing colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* American Society of Anesthesiologists (ASA) physical status classification I-III
* Preoperative Mini-Mental State Examination (MMSE) score > 23
* Patients scheduled for elective colorectal surgery under general anesthesia. Disease diagnoses include colorectal cancer, benign polyps, benign strictures, or diverticular disease.
* Provide informed consent

Exclusion Criteria:

* Presence of psychiatric disorders, cognitive impairment, or language communication barriers that may affect assessment compliance.
* Body Mass Index (BMI) ≥ 35 kg/m².
* Severe hepatic dysfunction (Child-Pugh Class C) or renal dysfunction (estimated glomerular filtration rate < 30 ml/min/1.73m² and/or receiving renal replacement therapy).
* Pre-existing severe gastrointestinal dysfunction (e.g., intestinal obstruction, active inflammatory bowel disease, severe constipation/diarrhea); receipt of neoadjuvant therapy preoperatively; planned stoma creation surgery; or scheduled for low rectal surgery (e.g., low anterior resection, abdominoperineal resection).
* History of neuromuscular disorders (e.g., myasthenia gravis) or malignant hyperthermia.
* History of opioid abuse, or chronic non-surgical pain requiring long-term analgesic therapy.
* Anticipated difficult airway, or patients planned for postoperative transfer to the intensive care unit (ICU) while intubated.
* Contraindications to the use of neostigmine, atropine, sugammadex, or rocuronium (e.g., known drug allergy, epilepsy, unstable angina, asthma, glaucoma, uncontrolled malignant arrhythmias especially atrioventricular block, severe cardiac valve stenosis); or current use of medications that may significantly influence the effects of neuromuscular blocking agents (e.g., antibiotics such as tetracyclines, aminoglycosides, polymyxins, and clindamycin; antiepileptic drugs; lithium; certain antidepressants such as sertraline and amitriptyline).
* Pregnant or lactating women.
* Current participation in other clinical trials that may interfere with the results of this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients recovering gastrointestinal function within 72 hours after surgery (assessed using the GI-3 criterion). | up to 72 hours after surgery
  GI-3 is defined as the ability to tolerate oral intake (no significant nausea or vomiting during three consecutive meals of solid food and beverages) and the passage of flatus or stool (whichever occurs first).

SECONDARY OUTCOMES:
Time to achieve GI-3 (hours) | up to 10 days after surgery
  Defined as the time from the end of anesthesia until the patient meets the GI-3 criteria.
Time to achieve GI-2 (hours) | up to 10 days after surgery
  GI-2 is defined as the ability to tolerate oral intake (no significant nausea or vomiting during three consecutive instances of eating and drinking) and having a bowel movement
Incidence of Prolonged Postoperative Ileus (PPOI) | 120 hours (5 days) after surgery
  Defined as the proportion of patients who fail to meet the GI-3 criteria by 120 hours (5 days) after surgery. Diagnosis requires radiographic imaging (e.g., abdominal X-ray or CT scan) to rule out mechanical obstruction, intra-abdominal infection, or other related complications (e.g., anastomotic leakage).
Time to first oral intake | Assessed up to 10 days after surgery
  record the time from surgery to first time of oral intake
Time to first passage of flatus | Assessed up to 10 days after surgery
  record the time from surgery to first time passage of flatus
Time to first defecation | Assessed up to 10 days after surgery
  record the time from surgery to first time defecation
Time to first ambulation | Assessed up to 10 days after surgery
  record the time from surgery to first time ambulation
Incidence of adverse events during the recovery period | Within 2 hours after extubation
  any adverse events such as hypoxia will be recorded within this 2hrs time frame
Intake, Feeling nausea, Emesis, physical Exam, and Duration of symptoms (I-FEED) score at 24, 48, and 72 hours after surgery | At 24, 48, and 72 hours after surgery
  The I-FEED scoring system incorporates five elements: intake (score: 0, 1, 3), feeling nauseated (score: 0, 1, 3), emesis (score: 0, 1, 3), results of physical exam (score: 0, 1, 3), and duration of symptoms (score: 0, 1, 2), with a total score ranging from 0 to 14. A higher score indicates poorer postoperative gastrointestinal recovery.
Visual Analog Scale (VAS) score at rest and during activity | At 24, 48, and 72 hours after surgery
  The VAS score ranges from 0 to 10, with a higher score indicating greater pain intensity
Total opioid consumption | Within 24, 48, and 72 hours after surgery
  the postoperative opioid comsumption will recorded in morphine equivalent dose.
Postoperative Nausea and Vomiting (PONV) | At 24, 48, and 72 hours after surgery
  PONV scores (range from 0-3, a higher score indicates that the patient is experiencing more severe and frequent symptoms of postoperative nausea and vomiting), number of vomiting episodes, and the use of rescue antiemetic medications (name and dose)
Postoperative Quality of Recovery | From postoperative day 1 to day 7 (or until discharge, whichever comes first)
  Assessed using the QoR-15 questionnaire preoperatively and daily
Incidence of postoperative delirium | Within 7 days after surgery (or until discharge, whichever comes first)
  Assessed using the Confusion Assessment Method (CAM)
Time to meet medically defined discharge criteria (days) | Assessed up to 30 days after surgery
  Defined as the time when the patient meets all of the following criteria: ability to independently consume fluids/nutrition, adequate pain control with oral analgesics, ability to ambulate independently, recovery of gastrointestinal function according to GI-3 criteria, and absence of medical contraindications.
Patient-assessed time to readiness for discharge (days) | Assessed up to 30 days after surgery
  Defined as the time when the patient meets the medically defined discharge criteria and subjectively agrees to be discharged.
Quality of life assessment using the European Quality of Life 5-Dimension 5-Level (EQ-5D-5L) questionnaire | Preoperatively, postoperative day 7, and postoperative day 30
  The EQ-5D-5L consists of 25 items (rated from 1 = best condition to 5 = worst condition) across five domains: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression, with a cumulative score ranging from 5 to 25. Higher EQ-5D-5L scores indicate poorer health status, reflecting greater difficulty in daily activities, higher levels of pain, or emotional distress. Conversely, lower scores indicate better health with fewer or no problems.
Postoperative length of hospital stay | From postoperative Day 1 to hospital discharge, assessed up to postoperative 30 days
  the time from surgery to hospital discharge
Total hospitalization costs | From hospital admission to hospital discharge, assessed up to postoperative 30 days
  in Chinese Yuan, RMB
Incidence of complications | Within 30 days after surgery
  All complications occurring within 30 days after surgery will be recorded and graded according to the Clavien-Dindo classification system
Days Alive and Out of Hospital within 30 days after surgery (DAOH30) | Within 30 days after surgery
  DAOH30 is defined as the number of days the patient is alive and not hospitalized in any medical facility (including rehabilitation institutions) within 30 days after surgery
Adverse events (AEs) | From the time the patient signs the informed consent form until the end of the study follow-up (30 days after surgery)
  Recorded any adverse event during the study peroid, no matter the AEs related to the intervention or not.